CLINICAL TRIAL: NCT02494895
Title: Ticagrelor Monotherapy After 3 Months in the Patients Treated With New Generation Sirolimus Stent for Acute Coronary Syndrome (TICO Study)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-2014-0066
Record Dates: First submitted 2015-07-07; First posted 2015-07-10 (Estimated); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ticagrelor monotherapy (Experimental): Ticagrelor monotherapy at 3 months after PCI
  Interventions: Drug: Ticagrelor monotherapy
- Ticagrelor with Aspirin (Active Comparator): Ticagrelor with Aspirin DAPT(Dual Anti-platelet Treatment)
  Interventions: Drug: Ticagrelor with Aspirin DAPT(dual antiplatelet treatment)

INTERVENTIONS:
Drug: Ticagrelor monotherapy — Ticagrelor (Brilinta®) is indicated for the prevention of thrombotic events (for example stroke or heart attack) in people with acute coronary syndrome or myocardial infarction with ST elevation. Patients will be randomized to stop aspirin at 3 months after PCI.
  Other Names: Brilinta®
  Arms: Ticagrelor monotherapy
Drug: Ticagrelor with Aspirin DAPT(dual antiplatelet treatment) — Ticagrelor (Brilinta®) is indicated for the prevention of thrombotic events (for example stroke or heart attack) in people with acute coronary syndrome or myocardial infarction with ST elevation. Patients will be randomized to continue DAPT (aspirin+ticagrelor) up to 1 year.
  Arms: Ticagrelor with Aspirin

SUMMARY:
To compare the clinical outcomes of dual antiplatelet therapy with aspirin and ticagrelor vs. ticagrelor monotherapy at 3 months after PCI in patients with acute coronary syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 19 years old
* Patients who received new generation sirolimus-eluting (Osiro®) stent implantation for treating ACS
* Patients without significant clinical events such as MI, stent thrombosis or revascularization until 3 months after PCI
* Provision of informed consent

Exclusion Criteria:

* Age > 80 years
* Increased risk of bleeding, anemia, thrombocytopenia
* A need for oral anticoagulation therapy
* Pregnant women or women with potential childbearing
* Life expectancy < 1 year
* Patients who treated with strong CYP3A4 inhibitors (e.g. ketoconazole, clarithromycin, nefazodone, ritonavir, or atazanavir)
* Patients who had history of intracranial hemorrhage
* Moderate to severe hepatic dysfunction
* Increased risk of bradycardia-related symptom (Guidance and reference)

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3056 (Estimated)
Dates: Start 2015-08-01 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular clinical events (MACCE) | 1 year after the procedure
major bleeding | 1 year after the procedure
  Major bleeding means 1) any intracranial bleeding (excluding microhemorrhages <10 mm evident only on gradient-echo MRI), 2) clinically overt signs of hemorrhage associated with a drop in hemoglobin of ≥5 g/dL or a ≥15% absolute decrease in haematocrit, and 3) fatal bleeding (bleeding that directly results in death within 7 days) in accordance with TIMI Bleeding Criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Department of Internal Medicine, Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Derived] Jin IT, Kim Y, Heo SJ, Lee YJ, Lee SJ, Hong SJ, Ahn CM, Kim JS, Cho DK, Ko YG, Choi D, Hong MK, Kim BK. Comparison of Short-term and Standard Duration Dual Antiplatelet Therapy in Elderly Patients: A Pooled Analysis of Five Korean Randomized Clinical Trials. Korean Circ J. 2025 Dec;55(12):1125-1137. doi: 10.4070/kcj.2025.0093. Epub 2025 Jul 14. PMID 41044734
- [Derived] Cho JY, Joo D, Yun KH, Kim BK, Hong MK, Jang Y, Oh SK. Clinical implication of ticagrelor monotherapy in patients with small vessel coronary artery disease: results from the TICO randomized trial. Front Cardiovasc Med. 2023 Aug 8;10:1237826. doi: 10.3389/fcvm.2023.1237826. eCollection 2023. PMID 37614943
- [Derived] Kim BG, Hong SJ, Kim BK, Lee YJ, Lee SJ, Ahn CM, Shin DH, Kim JS, Ko YG, Choi D, Hong MK, Jang Y. Body mass index affecting ticagrelor monotherapy vs. ticagrelor with aspirin in patients with acute coronary syndrome: A pre-specified sub-analysis of the TICO randomized trial. Front Cardiovasc Med. 2023 Mar 30;10:1128834. doi: 10.3389/fcvm.2023.1128834. eCollection 2023. PMID 37063970
- [Derived] Lee YJ, Suh Y, Kim JS, Cho YH, Yun KH, Kim YH, Cho JY, Her AY, Cho S, Jeon DW, Yoo SY, Cho DK, Hong BK, Kwon H, Hong SJ, Ahn CM, Shin DH, Nam CM, Kim BK, Ko YG, Choi D, Hong MK, Jang Y; TICO investigators. Ticagrelor Monotherapy After 3-Month Dual Antiplatelet Therapy in Acute Coronary Syndrome by High Bleeding Risk: The Subanalysis From the TICO Trial. Korean Circ J. 2022 Apr;52(4):324-337. doi: 10.4070/kcj.2021.0321. Epub 2021 Dec 28. PMID 35129317
- [Derived] Lee SJ, Lee YJ, Kim BK, Hong SJ, Ahn CM, Kim JS, Ko YG, Choi D, Hong MK, Jang Y. Ticagrelor Monotherapy Versus Ticagrelor With Aspirin in Acute Coronary Syndrome Patients With a High Risk of Ischemic Events. Circ Cardiovasc Interv. 2021 Aug;14(8):e010812. doi: 10.1161/CIRCINTERVENTIONS.121.010812. Epub 2021 Jul 20. PMID 34281363
- [Derived] Kim YH, Her AY, Kim BK, Hong SJ, Ahn CM, Kim JS, Ko YG, Choi D, Hong MK, Jang Y. Impact of preprocedural coronary flow grade on duration of dual antiplatelet therapy in acute myocardial infarction. Sci Rep. 2021 Jun 3;11(1):11735. doi: 10.1038/s41598-021-91130-5. PMID 34083627
- [Derived] Cho JY, Lee SY, Yun KH, Kim BK, Hong SJ, Ko JS, Rhee SJ, Oh SK, Shin DH, Ahn CM, Kim JS, Ko YG, Choi D, Hong MK, Jang Y. Factors Related to Major Bleeding After Ticagrelor Therapy: Results from the TICO Trial. J Am Heart Assoc. 2021 Apr 6;10(7):e019630. doi: 10.1161/JAHA.120.019630. Epub 2021 Mar 19. PMID 33739127
- [Derived] Lee SJ, Cho JY, Kim BK, Yun KH, Suh Y, Cho YH, Kim YH, Her AY, Cho S, Jeon DW, Yoo SY, Cho DK, Hong BK, Kwon HM, Hong SJ, Ahn CM, Shin DH, Nam CM, Kim JS, Ko YG, Choi D, Hong MK, Jang Y; TICO Investigators. Ticagrelor Monotherapy Versus Ticagrelor With Aspirin in Patients With ST-Segment Elevation Myocardial Infarction. JACC Cardiovasc Interv. 2021 Feb 22;14(4):431-440. doi: 10.1016/j.jcin.2020.11.036. PMID 33602439
- [Derived] Yun KH, Cho JY, Lee SY, Rhee SJ, Kim BK, Hong MK, Jang Y, Oh SK; TICO Investigators. Ischemic and Bleeding Events of Ticagrelor Monotherapy in Korean Patients With and Without Diabetes Mellitus: Insights From the TICO Trial. Front Pharmacol. 2021 Jan 14;11:620906. doi: 10.3389/fphar.2020.620906. eCollection 2020. PMID 33519487
- [Derived] Kim BK, Hong SJ, Cho YH, Yun KH, Kim YH, Suh Y, Cho JY, Her AY, Cho S, Jeon DW, Yoo SY, Cho DK, Hong BK, Kwon H, Ahn CM, Shin DH, Nam CM, Kim JS, Ko YG, Choi D, Hong MK, Jang Y; TICO Investigators. Effect of Ticagrelor Monotherapy vs Ticagrelor With Aspirin on Major Bleeding and Cardiovascular Events in Patients With Acute Coronary Syndrome: The TICO Randomized Clinical Trial. JAMA. 2020 Jun 16;323(23):2407-2416. doi: 10.1001/jama.2020.7580. PMID 32543684